CLINICAL TRIAL: NCT02197377
Title: Comparison of The Laryngeal Mask Airway Supreme™ Versus Unique™ in Edentulous Geriatric Patients
Brief Title: The Laryngeal Mask Airway in Edentulous Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Anaesthesiology and Reanimation, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 178/2009
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2017-12

CONDITIONS: Anaesthesia
Keywords: Laryngeal mask airway, edentulous geriatric patient

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group LMA Unique (Active Comparator): The supraglottic airway devices were deflated fully before insertion. Size 4 LMA was used for those with a weight of 50-70 kg and size 5 LMA for those between 70-100 kg. After insertion, each device was inflated with a hand-held airway manometer (Rusch, Germany) to an intracuff pressure of 60 cm H2O.The oropharyngeal leak pressure was determined by transiently stopping ventilation and closing the adjustable pressure-limiting valve with a fresh gas flow of 3 L/min until airway pressure reached a steady state and a voice of leakage was heard. The airway pressure was not allowed to exceed 40 cm H2O.
  Interventions: Device: Group LMA Unique™
- Group LMA Supreme (Experimental): The supraglottic airway devices were deflated fully before insertion. Size 4 LMA was used for those with a weight of 50-70 kg and size 5 LMA for those between 70-100 kg. After insertion, each device was inflated with a hand-held airway manometer (Rusch, Germany) to an intracuff pressure of 60 cm H2O.The oropharyngeal leak pressure was determined by transiently stopping ventilation and closing the adjustable pressure-limiting valve with a fresh gas flow of 3 L/min until airway pressure reached a steady state and a voice of leakage was heard. The airway pressure was not allowed to exceed 40 cm H2O.
  Interventions: Device: Group LMA Supreme™

INTERVENTIONS:
Device: Group LMA Unique™ — The supraglottic airway devices were deflated fully before insertion. After placement an effective airway was defined as the presence of normal thoracoabdominal movement and a square-wave end-tidal carbon dioxide trace.
  Other Names: Laryngeal Mask Airway Unique; LMA Unique (The Laryngeal Mask Company Limited, Singapore)
  Arms: Group LMA Unique
Device: Group LMA Supreme™ — The supraglottic airway devices were deflated fully before insertion.The supraglottic airway devices were deflated fully before insertion. After placement an effective airway was defined as the presence of normal thoracoabdominal movement and a square-wave end-tidal carbon dioxide trace.
  Other Names: Laryngeal Mask Airway Supreme; Teleflex, The Laryngeal Mask Company Limited, Singapore
  Arms: Group LMA Supreme

SUMMARY:
With an aging population a prevalence of edentulous patients increased above 60 % among individuals aged ≥65 yr. Face mask ventilation of these edentulous patients is often difficult because of the inadequate fitting of the standard mask to the face. In addition, because of a reduction in muscle tone under general anesthesia, the air space in the oropharynx is reduced, and posterior displacement of the tongue, soft palate and epiglottis tend to close the airway. The laryngeal mask airway (LMA) provides a better alternative to the standard face mask if the facial contours of the patient are not suited to the standard face mask. It is more difficult to perform bag-mask ventilation in edentulous patients than in patients with intact dentition. The laryngeal mask airway (LMA) provides a better alternative to the standard face mask if the facial contours of the patient are not suited to the standard face mask.

We aimed to compare the routinely used laryngeal mask airway in our clinic, the LMA Unique™ with the newly released LMA Supreme™ in edentulous elderly patients for the success in first attempt insertion, ease and time of insertion, and oropharyngeal leak pressure.

DETAILED DESCRIPTION:
After Ethical Committee approval and written informed consent were obtained, sixty edentulous patients (American Society of Anesthesiologists physical status (ASA) grade I-III, aged over 65 years) undergoing elective surgery were included into the study. Patients with dentures had to remove their dentures before surgery at the ward. The supraglottic airway device was inserted into each patient in a random order. A statistician independent of the clinical investigators generated the randomization sequence using a computerized program. Patients were excluded if they had a known or predicted difficult airway, a body mass index > 35 kg/m2, or were at risk of aspiration. All cases were conducted by anesthetists who had experience over 5 years of LMA insertion.

Demographic parameters, Mallampati classification and the duration of surgery were recorded. Patients were routinely monitored using ECG, non-invasive blood pressure measurement, pulse oximetry and end-tidal carbon dioxide tension. Depth of anesthesia was monitored with bispectral index (BIS).

Patients were premedicated with midazolam 0.02 mg/kg when venous access was obtained. After 3 min preoxygenation with 100 % oxygen via face mask, anesthesia was induced with fentanyl 1-2 µg/kg and propofol 1-2 mg/kg. When the BIS value was 40-60 the predetermined supraglottic airway device was inserted according to the manufacturer's recommendations. The supraglottic airway devices were deflated fully before insertion. Size 4 LMA was used for those with a weight of 50-70 kg and size 5 LMA for those between 70-100 kg. After insertion, each device was inflated with a hand-held airway manometer (Rusch, Germany) to an intracuff pressure of 60 cm H2O.

An effective airway was defined as the presence of normal thoracoabdominal movement and a square-wave end-tidal carbon dioxide trace. General anesthesia was maintained with sevoflurane, O2 and N2O.

Insertion time was defined as the time from picking up the airway device until connection to the airway circuit. Ease of insertion was graded by the attending anesthesiologist as easy, fair or difficult. If after three attempts insertion was still not successful, the other device was used. If insertion of the other device also failed the patient was endotracheally intubated.

Before the oropharyngeal leak test was carried out, the face of the patient was covered so that the observer was blinded to the airway device. The oropharyngeal leak pressure was determined by transiently stopping ventilation and closing the adjustable pressure-limiting valve with a fresh gas flow of 3 L/min until airway pressure reached a steady state and a voice of leakage was heard. The airway pressure was not allowed to exceed 40 cm H2O.

After successful placement of the LMA Supreme™, a 12 French gauge gastric catheter was inserted via the gastric channel.

Any episode of hypoxemia (SpO2 < 90%), aspiration or regurgitation,bronchospasm and airway obstruction were documented. After removal of the LMA, it was examined for the presence of visible blood.

In the postanesthesia care unit, a research assistant, who was blinded to the group allocation, interviewed the patients using a predetermined questionnaire to collect data on the postoperative pharyngolaryngeal adverse events. The presence or absence of sore throat, dysphonia and dysphagia was assessed at 1 and 24 h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* 65 years and older

Exclusion Criteria:

* Any neck or upper respiratory pathology
* Those at risk of gastric content regurgitation/aspiration (previous upper gastro-intestina system surgery, known hiatus hernia, gastroesophageal reflux, history of peptic ulcer, full stomach, pregnancy)
* Possibility of and those with history of difficult intubation (history of impossible intubation, Mallampati classification 3-4, sterno mental distance less than 12 cm, thyromental distance less than 6 cm, head extension less than 90 degrees, mouth opening less than 1.5 cm)
* Those with low pulmonary compliance or high airway resistance (morbid obesity, lung disease)
* Throat pain, dysphagia and dysphonia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TANGUL KILIÇ, M.D., Principal Investigator — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation; SEMİH KUCUKGUCLU, M.D., Study Director — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation, Izmi̇r, Narlıdere, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group LMA Unique: The supraglottic airway devices were deflated fully before insertion. Size 4 LMA was used for those with a weight of 50-70 kg and size 5 LMA for those between 70-100 kg. After insertion, each device was inflated with a hand-held airway manometer (Rusch, Germany) to an intracuff pressure of 60 cm H2O.
  Group LMA Supreme™: The supraglottic airway devices were deflated fully before insertion.
- Group LMA Supreme: The supraglottic airway devices were deflated fully before insertion. Size 4 LMA was used for those with a weight of 50-70 kg and size 5 LMA for those between 70-100 kg. After insertion, each device was inflated with a hand-held airway manometer (Rusch, Germany) to an intracuff pressure of 60 cm H2O.
  Group LMA Unique™: The supraglottic airway devices were deflated fully before insertion.
Period: Overall Study
Arm/Group | Group LMA Unique | Group LMA Supreme
Started | 30 | 30
Completed | 30 | 27
Not Completed | 0 | 3
Not completed — Insertion Failure | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group LMA Unique | Group LMA Supreme | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 27 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 21 | 16 | 37
Region of Enrollment [Number; unit: participants] — Three patients LMA supreme insertion failure occurred and these patients were excluded from further analysis.
  participants
    Turkey | 30 | 27 | 57

OUTCOME MEASURES:

1. Primary Outcome: First Attempt's Success Rate of Insertion
Description: Edentulous elderly patients for the success in first attempt insertion, ease and time of insertion (second).
Time Frame: after anaesthesia induction
Population: Non parametric data between groups were analyzed with the X2-test, while parametric data were compared with unpaired t-test. P < 0.05 was considered significant. 3 LMA insertion failed in Group LMA Supreme. Total 27 patients included analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Group LMA Unique | Group LMA Supreme
Number analyzed (Participants) | 30 | 27
percentage of participants | 73.3 | 86.6

2. Secondary Outcome: Oropharyngeal Leak Pressure
Description: The aim of this study is to compare on the oropharyngeal leak pressure in LMA Unique™ and LMA Supreme™ applications
Time Frame: before surgery
Population: Non parametric data between groups were analyzed with the X2-test, while parametric data were compared with unpaired t-test. P < 0.05 was considered significant.
Measure: Mean (Standard Deviation); unit: cm H20
Arm/Group | Group LMA Unique | Group LMA Supreme
Number analyzed (Participants) | 30 | 27
cm H20 | 17.1 (6.33) | 20.56 (8.22)

ADVERSE EVENTS:
Arm/Group | Group LMA Unique | Group LMA Supreme
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/27
Other Adverse Events (participants affected / at risk) | 0/30 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No